CLINICAL TRIAL: NCT00488384
Title: Acitretin Plasma Levels Under Hemodialysis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of subjects
Sponsor: Günther Hofbauer (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Günther Hofbauer, senior staff physician, University of Zurich
Organization: University of Zurich (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007DR2065 EK674
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Squamous cell carcinoma of the skin under hemodialysis
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Acitretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- a (Other): single arm only. Only open label treatment anticipated
  Interventions: Drug: Chemopreventive application (Acitretin)

INTERVENTIONS:
Drug: Chemopreventive application (Acitretin) — Chemopreventive application (Acitretin)

SUMMARY:
Acitretin is given to hemodialysis patients who have developed in-situ or invasive squamous cell carcinoma of the skin in increasing doses up to 25 mg daily for one year.

DETAILED DESCRIPTION:
Acitretin is given to hemodialysis patients who have developed in-situ or invasive squamous cell carcinoma of the skin in increasing doses up to 25 mg daily for one year. Plasma levels of acitretin will be monitored and influence of hemodialysis on acitretin plasma levels will be determined. Number of in-situ or invasive squamous cell carcinoma of the skin cases will be determined.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Hemodialyis patients with at least one case of in-situ or invasive squamous cell carcinoma of the skin

Exclusion criteria:

* Hepatopathy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Plasma levels acitretin | 2009

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Clinic for Dermatology University Hospital of Zurich, Zurich, Switzerland